CLINICAL TRIAL: NCT07293013
Title: A Study on the Effectiveness of Olive Oil Mouthwash in Alleviating Chemoradiotherapy-induced Oral Mucositis in Patients With Head and Neck Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB2022100
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis in Head and Neck Cancer; Chemo-radiotherapy
Keywords: Oral Mucositis; Head and Neck Cancer; Chemo-radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: Participants were recruited from the outpatient radiology department of a hospital in southern Taiwan. This study employed a randomized controlled trial (RCT) design in accordance with the research objectives. Microsoft Excel was used to perform random allocation, evenly assigning participants to either the experimental group or the control group. Matching was conducted based on age and cancer type to minimize differences in baseline characteristics between the two groups.
Who Masked: Outcomes Assessor
Masking Description: The severity of oral mucositis (OM) was assessed independently by two evaluators. The first evaluator, a physician, conducted direct clinical assessments of the patients' oral mucosa using the Radiation Therapy Oncology Group (RTOG) grading scale. The second evaluator, a hematology-oncology nurse, evaluated de-identified photographs of the patients' oral mucosa. These photographs were taken by the researcher using a specialized intraoral camera. Both evaluators performed the assessments independently and were blinded to the participants' group allocation to ensure objectivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olive oil mouthwash (Experimental)
  Interventions: Other: olive oil mouthwash
- Standard care (No Intervention)

INTERVENTIONS:
Other: olive oil mouthwash — . The procedures and timing of the olive oil mouth rinse were as follows:
  A volume of 10 mL of olive oil was held in the mouth and used for rinsing for 2 minutes. Participants were instructed not to tilt their heads backward during rinsing to prevent choking.
  At home, the olive oil mouth rinse was performed as the final step of routine oral hygiene. If an antimicrobial mouthwash had been prescribed by the physician, it was used prior to the olive oil rinse.
  The olive oil mouth rinse intervention was initiated on the first day of radiotherapy or concurrent chemoradiotherapy (CCRT) and continued until completion of radiotherapy.
  Participants were instructed to refrain from eating or drinking for 30 minutes after each olive oil mouth rinse.
  Arms: olive oil mouthwash

SUMMARY:
Backgroud: Radiation therapy and concurrent chemoradiotherapy are the main treatment methods for patients with head and neck cancer, which often lead to many severe oral mucositis (OM). It is easy to cause dry mouth and infection, which seriously affects the comfort and quality of life of patients. There are many pharmacological and non-pharmacological mouthwash solutions in clinical practice, the purpose of which is to reduce bacterial accumulation in order to prevent and improve OM. Olive oil has powerful moisturizing, antioxidant and anti-inflammatory properties. There is no research on the use of olive oil in the prevention or treatment of OM.

Objective: The purpose of this study was to evaluate the preventive and therapeutic effects of olive oil as a mouthwash solution on OM caused by radiation therapy or concurrent chemoradiotherapy.

Methods: The research design of this study is a randomized controlled trial. Patients from a radiation oncology clinic of a regional teaching hospital in southern China were invited to participate in the study by intentional sampling. The study will be followed for 12 weeks and will collect data before and after treatment with olive oil mouthwash or standard care. Assessment tools include demographic characteristics, severity of OM (RTOG and OMAS), degree of dry mouth (XQ and Saxon test), pain severity(VAS), Shortened General Comfort Questionnaire (SGCQ) and head and neck cancer patients quality of life scale (FACT-H&N). The research data will be statistically analyzed by SPSS 22.0 statistical software, and the statistical significance is defined as the P value less than 0.05 as the significant level. Statistical methods include 1) Descriptive statistics include times, percentages, averages, standard deviations, etc. 2) Inferential statistics: Chi-square test, independent t-test, paired t-test and Logistic regression were used to compare the post-test data between the experimental group and the control group, and to detect the effectiveness of intervention measures and 3) Using generalized estimating equations (GEE) to predict the effect of interventions (repeated measures) on OM severity, dry mouth, body weight, quality of life and comfort scores.

Expected outcomes: This study aimed to investigate the efficacy of gargling with olive oil in reducing the incidence of OM, severity of OM, severity of dry mouth, severity of pain, and improved patient comfort and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* A. Aged 20 years or older. B. Diagnosed with a primary cancer located in the head and neck region and preparing to undergo radiotherapy or concurrent chemoradiotherapy (CCRT). For the purposes of this study, CCRT is defined as receiving chemotherapy within one week before or after the first day of radiotherapy.

C. The total prescribed radiotherapy dose is between 6000 and 7200 cGy. D. Conscious and able to communicate in Mandarin or Taiwanese. E. Willing to participate in the study after receiving an explanation, and capable of signing the informed consent form.

Exclusion Criteria:

A. Patients diagnosed with recurrent head and neck cancer undergoing a second course of radiotherapy or CCRT.

B. Patients who are allergic or have a history of allergy to any component of the intervention used in this study.

C. Patients who are unable to open their mouth due to skin grafting. D. Patients with known metastasis (M1). E. Patients who have already developed oral mucositis (OM). F. Patients with skin diseases, autoimmune disorders, or those deemed unsuitable for the study by the physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment severity of OM | 12 Weeks
  The study will be followed for 12 weeks and will collect data before and after treatment with olive oil mouthwash or standard care. Assessment tools include demographic characteristics, severity of OM (RTOG and OMAS)

SECONDARY OUTCOMES:
degree of dry mouth | 12 weeks
  Assessment tools include XQ and Saxon test
pain severity | 12 Weeks
  Assessment tools VAS
General Comfort | 12 Weeks
  Assessment tools Shortened General Comfort Questionnaire (SGCQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Chia-Yi City, Taiwan

IPD SHARING:
Plan to Share IPD: No